CLINICAL TRIAL: NCT02155556
Title: Diurnal Changes of the Cornea - a Pilot Study
Status: Completed | Type: Observational
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, MD, MBA, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Other Study IDs: DIU
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy volunteers

SUMMARY:
Aim of this study is to gain a better understanding of the diurnal changes of the cornea to improve toric IOL power calculations.

DETAILED DESCRIPTION:
Higher patient expectations concerning unaided visual acuity after cataract surgery has led to an increase in use of toric intraocular lenses (toric IOLs) for the correction of corneal astigmatism. Although it was shown that toric IOLs significantly reduce astigmatism, there is still some difficulty in predicting the remaining astigmatism correctly. The main source of error appears to be the pre-operative measurement of the cornea. However, it is questionable, if this error derives from a measurement error due to the imprecise measurement technique, or natural diurnal changes of the cornea. Additionally, measurements of the cornea pose several challenges: different corneal biometry devices cannot be used interchangeably and it is difficult to decide, which device is measuring the cornea correctly as there is no gold standard.

Especially, in eyes with small corneal astigmatism the error increases. Recently it was shown that the astigmatism meridian was on median 9° off for corneas with 1.0D of astigmatism and only 4° for corneas with 2.0D of astigmatism. Similar findings were observed by Shammas et al. Norrby furthermore showed that 5% of all corneas show more than 0.5D of fluctuations between measurements at different (post-operative) time-points. The reasons are not explored, but diurnal changes, temperature and humidity potentially influencing the tear film, as well as pupil size and asphericity of the cornea could play a role. Read and Collins observed diurnal changes of corneal radii within 24 hours, but in their study only young healthy volunteers were included and only one measurement device (Scheimpflug imaging, Pentacam HR) was used. Lau and Pye and Shen et al. measured the diurnal changes of the cornea, but no data concerning corneal radii were reported. Harper et al. observed diurnal changes of the central corneal thickness. However, none of these studies investigated on diurnal changes of the corneal radii in the elderly population. Aim of this study is to gain a better understanding of the diurnal changes of the cornea to improve toric IOL power calculations.

ELIGIBILITY:
Inclusion Criteria:

* 21 years, or above
* Signed informed consent

Exclusion Criteria:

* Ophthalmic diseases such as significant macular degeneration, glaucoma, diabetic retinopathy, etc.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 volunteers/patients (10 patients >50 years old; 5 patients with a corneal astigmatism of >1 D)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Descriptive analysis of diurnal changes of the corneal radii (in diopters) and orientation of the steep meridian (in degrees) in young healthy subjects and elderly patients | 24 hours

SECONDARY OUTCOMES:
Comparison of the corneal radii (in diopters) and orientation of the steep meridian (in degrees) between different measuring devices | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, MBA, Principal Investigator — VIROS - Vienna Institute for Research in Ocular Surgers - Departement of Opthalmology - Hanusch Hospital Vienna, Vienna, Austria 1140
Locations (1):
- VIROS - Vienna Institute for Research in Ocular Surgers - Departement of Opthalmology - Hanusch Hospital, Vienna, Austria